CLINICAL TRIAL: NCT03297970
Title: Bogota School Children Cohort
Acronym: BoSCCo
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Universidad de la Sabana (Other); Foundation for Research in Nutrition and Health (FINUSAD) (Unknown)
Responsible Party: Principal Investigator, Eduardo Villamor, Professor, University of Michigan
Other Study IDs: HUM00043252
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Nutrition; Child Health; Child Growth; Neurocognitive Development; Sexual Maturation; Infectious Morbidity; Behavior Problem
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma, serum, and DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bogota School Children Cohort: Children are classified according to exposure levels of:
  Micronutrient biomarker indicators:
  * Ferritin
  * Hemoglobin
  * Mean corpuscular volume
  * Zinc
  * Vitamin A
  * Vitamin B12
  * Folate
  * Vitamin D
  Serum fatty acids
  Inflammatory biomarkers:
  * C-reactive protein
  Diet
  Socioeconomic status indicators
  Anthropometric indicators
  Incidence of infectious morbidity symptoms
  DNA biomarkers

SUMMARY:
This observational study investigates the associations of nutritional indicators, biomarkers, sociodemographic conditions, and infections with child health, as well as physical, behavioral, and cognitive development. Investigators recruited a random sample of 3202 children from primary public schools in Bogota, Colombia in February 2006 and followed them for a median of 6.5 years. Investigators hypothesized that poor nutritional status at the time of recruitment in middle childhood would be related to adverse health outcomes through adolescence.

ELIGIBILITY:
Inclusion Criteria:

* Primary public school enrollment in February 2006

Exclusion Criteria:

* None

Ages: 5 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: Children were selected from primary public schools in Bogota, Colombia.
Sampling Method: Probability Sample
Enrollment: 3202 (Actual)
Dates: Start 2006-02-01 (Actual); Primary Completion 2015-08-11 (Actual); Study Completion 2015-08-11 (Actual)

PRIMARY OUTCOMES:
Externalizing behavior problems | Assessed at one point in time when the children were 11-18 years old.
  Adolescent behavior problems were ascertained with the Youth Self Report (YSR) questionnaire. The YSR is a self-administered questionnaire consisting of 112 statements addressing behaviors or feelings that adolescents rate as false, sometimes true, or very/often true. From responses to these questions, an Assessment Data Manager (ADM) software calculates continuous scores for aggressive behavior and rule breaking behavior. The sum of the aggressive and rule breaking behavior subscale scores constitute the total externalizing problems score.
Internalizing behavior problems | Assessed at one point in time when the children were 11-18 years old.
  Adolescent behavior problems were ascertained with the Youth Self Report (YSR) questionnaire. The sum of the anxious/depressed, withdrawn/depressed, and somatic complaint subscale scores constitute the total internalizing problems score.

SECONDARY OUTCOMES:
Behavior problem subscale scores (aggressive behavior, rule breaking behavior, anxious/depressed, withdrawn/depressed, somatic complaints, attention problems, social problems, and thought problems) | Assessed at one point in time when the children were 11-18 years old.
  Adolescent behavior problems were ascertained with the Youth Self Report (YSR) questionnaire.

OTHER OUTCOMES:
Body mass index change | Median 6.5 years from recruitment
  Change in body mass index for age Z-score from baseline to the last follow-up visit
Linear growth | Median 6.5 years from recruitment
  Change in height for age Z-score from baseline to the last follow-up visit
Age at menarche | Median 6.5 years from recruitment
  Reported age at first menstrual period
Grade repetition | 5 years
  Outcome of school grades between 2006-2011
Blood pressure | Median 6.5 years from recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Villamor, MD MPH DrPH, Principal Investigator — University of Michigan
Locations (2):
- Colombia (2):
  - FINUSAD - Foundation for Research in Nutrition and Health, Bogotá
  - University of La Sabana, Chía

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Robinson SL, Marin C, Oliveros H, Mora-Plazas M, Richards BJ, Lozoff B, Villamor E. Iron Deficiency, Anemia, and Low Vitamin B-12 Serostatus in Middle Childhood Are Associated with Behavior Problems in Adolescent Boys: Results from the Bogota School Children Cohort. J Nutr. 2018 May 1;148(5):760-770. doi: 10.1093/jn/nxy029. PMID 29897579